CLINICAL TRIAL: NCT01593527
Title: A Randomized Double-blind Active-controlled Trial of Canakinumab Versus Triamcinolone Acetonide on Reducing the Proportion of Patients With Any New Gouty Arthritis Flare(s) in Patients With Chronic Kidney Disease
Brief Title: Canakinumab in the Treatment of Gouty Arthritis Flare(s) and Prevention of New Flares in Patients With Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885H2402; 2011-001766-18 (EudraCT Number)
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2013-08

CONDITIONS: Acute Gouty Arthritis
Keywords: Frequent flares; Frequent attacks; gout; gouty arthritis; Chronic kidney disease; renal impairment; Anti-interleukin-1β monoclonal antibody; anti-inflammatory therapy
MeSH Terms: conditions — Gout; Arthritis, Gouty; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental): Canakinumab 150 mg s.c.
  Interventions: Drug: ACZ885
- Arm 2 (Experimental): Triamcinelone acetonide 40 mg i.m.
  Interventions: Drug: Triamcinelone acetonide

INTERVENTIONS:
Drug: ACZ885 — Canakinumab 150 mg s.c.
  Arms: Arm 1
Drug: Triamcinelone acetonide — Triamcinelone acetonide 40 mg i.m.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to confirm the efficacy and safety results obtained in a chronic kidney disease (CKD) subgroup of patients participating in Phase III studies in a larger, independent patient population with difficult to treat gouty arthritis and moderate to severe CKD (stage 3 - 4).

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of gouty arthritis History of ≥ 3 gouty arthritis flares within the previous 12 months
* Confirmed diagnosis/ documented history of chronic kidney disease (CKD) Stages 3or4
* Onset of current acute gouty arthritis flare within 3 days prior to randomization

Exclusion criteria:

* Hemodialysis CKD Stage 5 Organ transplantation
* Rheumatoid arthritis, evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis
* Live vaccinations within 3 months prior to randomization Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing new gouty arthritis flares during 12-week follow-up from dosing | 12 Weeks

SECONDARY OUTCOMES:
The time to the first new gout flare | 12 Weeks
Score on Visual Analog Scale at 72 hours to measure gouty arthritis pain intensity and resolution | 12 weeks
Number of patients needing rescue medication use during acute gouty arthritis flare(s) | 12 Weeks
Measurement of efficacy using inflammatory markers | 12 Weeks
Time to 50% reduction of baseline pain intensity in the most affected joint | 12 weeks